CLINICAL TRIAL: NCT01923168
Title: A Phase II Randomized, Double-blind Placebo Controlled, Study of Letrozole With or Without BYL719 or Buparlisib, for the Neoadjuvant Treatment of Postmenopausal Women With Hormone Receptor-positive HER2-negative Breast Cancer
Brief Title: Study of Letrozole With or Without BYL719 or Buparlisib, for the Neoadjuvant Treatment of Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBYL719A2201; 2013-001862-41 (EudraCT Number)
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: BYL719; alpelisib; Breast Cancer; BKM120; buparlisib; Pathological Complete Response; neoadjuvant; hormone receptor-positive; HER2 negative; Objective Response Rate
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib; NVP-BKM120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Alpelisib + Letrozole (Experimental): Participants took alpelisib 300 mg once daily plus letrozole 2.5 mg once daily.
  Interventions: Drug: alpelisib
- Buparlisib + Letrozole (Experimental): Participants took buparlisib 100 mg once daily or 5 days on/2 days off plus letrozole 2.5 mg once daily.
  Interventions: Drug: buparlisib
- Placebo + Letrozole (Placebo Comparator): Participants took matching Placebo (of alpelisib 300 mg once daily/buparlisib 100 mg once daily or 5 days on/2 days off) plus Letrozole 2.5 mg once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: alpelisib — BYL719 + Letrozole
  Other Names: BYL719
  Arms: Alpelisib + Letrozole
Drug: buparlisib — BKM120 + Letrozole
  Other Names: BKM120
  Arms: Buparlisib + Letrozole
Drug: Placebo — Placebo (of BYL719 or BKM120) + Letrozole
  Other Names: BYL719 Placebo, BKM120 Placebo
  Arms: Placebo + Letrozole

SUMMARY:
The purpose of the study was to determine whether treatment with a PI3K inhibitor plus letrozole led to an increase in pathologic clinical response and Objective Response Rate compared to treatment with placebo plus letrozole in patients with Breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult, female ≥ 18 years old at the time of informed consent
2. Patient has a histologically and/or cytologically confirmed diagnosis of breast cancer
3. Patient is postmenopausal.
4. Patient has T1c-T3, any N, M0, operable breast cancer
5. Patients must have measurable disease
6. Patient has diagnostic biopsy available for the analysis of PIK3CA mutation and Ki67 level.
7. Patient has estrogen-receptor and/or progesterone positive breast cancer as per local laboratory testing
8. Patient has HER2 negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0 or 1+ as per local laboratory testing

Exclusion Criteria:

1. Patient has locally recurrent or metastatic disease
2. Patient has received any systemic therapy (e.g. chemotherapy, targeted therapy, immunotherapy) or radiotherapy for current breast cancer disease before randomization.
3. Patient with type 1 diabetes mellitus or not adequately controlled type 2 diabetes mellitus
4. History of acute pancreatitis within 1 year of study entry
5. Uncontrolled hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (82):
- United States (23):
  - University of Alabama at Birmingham/ Kirklin Clinic Univ AL - PI, Birmingham, Alabama
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Los Angeles Hematology/Oncology Medical Group Onc Dept., Los Angeles, California
  - University of California at Los Angeles UCLA SC, Los Angeles, California
  - University of California San Francisco BYL719A2201 - SC, San Francisco, California
  - Emory University School of Medicine/Winship Cancer Institute SC, Atlanta, Georgia
  - Mercy Medical Center Medical Oncology & Hematology, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center/Johns Hopkins Med. Johns Hopkins Med. BYL719A2201, Baltimore, Maryland
  - Dana Farber Cancer Institute BYL719A2201, Boston, Massachusetts
  - Mayo Clinic - Rochester BYL719A2201 - SC, Rochester, Minnesota
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center Duke University Medical Center, Durham, North Carolina
  - Northwest Cancer Specialists Vancouver Loc, Portland, Oregon
  - Vanderbilt Ingram Cancer Center Vanderbilt Health 100 Oaks, Nashville, Tennessee
  - Texas Oncology, P.A., Bedford, Texas
  - Presbyterian Hospital of Dallas TexasOncology@PresbyterianHosp, Dallas, Texas
  - Texas Oncology Texas Oncology - Sammons, Dallas, Texas
  - Texas Oncology Houston Memorial City SC, Houston, Texas
  - Cancer Care Centers of South Texas HOAST CCC of So. TX- San Antonio(2), San Antonio, Texas
  - Cancer Therapy & Research Center UT Health Science Center InstituteForDrugDevelopment(5), San Antonio, Texas
  - Virginia Oncology Associates SC, Norfolk, Virginia
  - Seattle Cancer Care Alliance SC-3, Seattle, Washington
  - Northwest Medical Specialties Dept.ofNW Med. Specialties, Tacoma, Washington
- Novartis Investigative Site, Kingswood, New South Wales, Australia
- Austria (7):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Dornbirn, Vorarlberg
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Rankweil
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
  - Novartis Investigative Site, Villach
- Belgium (3):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Sint-Niklaas
- Brazil (4):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (3):
  - Novartis Investigative Site, Shumen
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Colombia (2):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bogotá
- Czechia (2):
  - Novartis Investigative Site, Olomouc, CZE
  - Novartis Investigative Site, Prague
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Kiel
- Novartis Investigative Site, Hong Kong SAR, Hong Kong
- Israel (3):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Japan (6):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Koto-ku, Tokyo
  - Novartis Investigative Site, Niigata
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Netherlands (4):
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Tilburg
- Spain (7):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mayer IA, Prat A, Egle D, Blau S, Fidalgo JAP, Gnant M, Fasching PA, Colleoni M, Wolff AC, Winer EP, Singer CF, Hurvitz S, Estevez LG, van Dam PA, Kummel S, Mundhenke C, Holmes F, Babbar N, Charbonnier L, Diaz-Padilla I, Vogl FD, Sellami D, Arteaga CL. A Phase II Randomized Study of Neoadjuvant Letrozole Plus Alpelisib for Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Breast Cancer (NEO-ORB). Clin Cancer Res. 2019 May 15;25(10):2975-2987. doi: 10.1158/1078-0432.CCR-18-3160. Epub 2019 Feb 5. PMID 30723140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of approximately 320 patients were planned to be randomized: this was based on 60 patients per arm in each cohort (PIK3CA mutant and PIK3CA wild-type) for the alpelisib+letrozole and placebo+letrozole arms, plus the estimated number of patients randomized to buparlisib+letrozole arm at the time this arm was discontinued.
Period: Overall Study
Arm/Group | Alpelisib + Letrozole | Buparlisib + Letrozole | Placebo + Letrozole
Started | 131 | 83 | 126
Completed | 94 | 44 | 109
Not Completed | 37 | 39 | 17
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Subject/guardian decision | 14 | 14 | 4
Not completed — Adverse Event | 12 | 12 | 0
Not completed — Physician Decision | 6 | 9 | 5
Not completed — Progressive disease | 4 | 3 | 7
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised all randomized subjects in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpelisib + Letrozole | Buparlisib + Letrozole | Placebo + Letrozole | Total
Number analyzed (Participants) | 131 | 83 | 126 | 340
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.53) | 65.2 (8.61) | 63.1 (8.31) | 64.1 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 83 | 126 | 340
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 117 | 68 | 105 | 290
  Asian | 7 | 4 | 10 | 21
  Black or African American | 3 | 3 | 5 | 11
  Other | 3 | 6 | 3 | 12
  Unknown | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Per Investigator Assessment for Alpelisib vs. Placebo for PIK3CA Mutant Cohort
Description: Pathologic complete response (pCR) defined as absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes following completion of 24 weeks of treatment by local assessment (ypT0/Tis ypN0). Patients who experienced progression of disease while undergoing neoadjuvant therapy, or who did not receive surgery for any reason, or received antineoplastic treatment other than study drug(s) before surgery were considered as non-responders for the calculation of pCR rate.
Time Frame: After 24 weeks of treatment
Population: The Full Analysis Set (FAS) for the PIK3CA mutant cohort comprised all randomized participants who were assigned to the PIK3CA mutant cohort based on tumor tissue for the randomization.
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 60 | 67
Percentage of Participants | 1.7 [0.2 to 6.3] | 3.0 [0.8 to 7.7]
Statistical Analysis 1: Comparison: Alpelisib + Letrozole vs Placebo + Letrozole; Test type: Other — Bayesian double criteria; p = 0.282, Posterior mean diff. & credible interval; Mean Difference (Final Values) = -1.3, 80% CI 2-sided [-4.5 to 1.7]

2. Primary Outcome: Pathological Complete Response (pCR) Per Investigator Assessment for Alpelisib vs. Placebo for PIK3CA Wild-type Cohort
Description: as for outcome 1
Time Frame: After 24 weeks of treatment
Population: The Full Analysis Set (FAS) for the PIK3CA wild-type cohort comprised all randomized participants who were assigned to the PIK3CA wild-type cohort based on tumor tissue for the randomization.
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 71 | 59
Percentage of Participants | 2.8 [0.8 to 7.3] | 1.7 [0.2 to 6.4]
Statistical Analysis 1: Comparison: Alpelisib + Letrozole vs Placebo + Letrozole; Test type: Other — Bayesian double criteria; p = 0.697, Posterior mean difference; Posterior mean difference; Mean Difference (Final Values) = 1.1, 80% CI 2-sided [-1.9 to 4.2]

3. Primary Outcome: Objective Response Rate Per Investigator Assessment According to RECIST 1.1 for Alpelisib vs. Placebo - PIK3CA Mutant Cohort
Description: Objective Response Rate (ORR) defined as the proportion of patients with a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) based on local investigator's assessment according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST) 1.1.
  BOR was assessed per MRI or Ultrasound and defined as per RECIST 1.1 as CR for a disappearance of all non-nodal target lesions (TL)/non-target lesions (NTL) and a reduction in short axis to < 10 mm of any pathological lymph nodes assigned as TL/NTL and no new lesion; as PR if not qualifying for CR but with a decrease from baseline ≥ 30% in the sum of diameter of all TL, no progression of NTL and no new lesion.
Time Frame: After 24 weeks of treatment
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 60 | 67
Percentage of Participants | 43.3 [34.6 to 52.4] | 44.8 [36.5 to 53.3]
Statistical Analysis 1: Comparison: Alpelisib + Letrozole vs Placebo + Letrozole; Test type: Other — Bayesian double criteria; p = 0.435, Posterior mean diff. & credible interval; Mean Difference (Final Values) = -1.4, 80% CI 2-sided [-12.5 to 9.7]

4. Primary Outcome: Objective Response Rate According to RECIST 1.1 Per Investigator Assessment for Alpelisib vs. Placebo - PIK3CA Wild-type Cohort
Description: as for outcome 3
Time Frame: After 24 weeks of treatment
Population: as for outcome 2
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 71 | 59
Percentage of Participants | 63.4 [55.1 to 71.0] | 61.0 [51.8 to 69.6]
Statistical Analysis 1: Comparison: Alpelisib + Letrozole vs Placebo + Letrozole; Test type: Other — Bayesian double criteria; p = 0.611, Posterior mean diff. & credible interval; Mean Difference (Final Values) = 2.4, 80% CI 2-sided [-8.4 to 13.2]

5. Secondary Outcome: pCR and Objective Response Rate According to RECIST 1.1 Criteria Per Investigator Assessment for Alpelisib vs. Placebo in PIK3CA Mutant Cohort Based on ctDNA
Description: pCR and Objective response rate according to RECIST 1.1 per investigator assessment after 24 weeks of treatment
Time Frame: After 24 weeks of treatment
Population: The FAS comprised all randomized participants. This analysis was to be done in patients with PIK3CA mutation based on Circulating tumor DNA (ctDNA). Data could not be reported as the ctDNA analysis was not done after the primary endpoint was negative.
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: pCR and Objective Response Rate According to RECIST 1.1 Criteria Per Investigator Assessment for Alpelisib vs. Placebo in PIK3CA Wild-type Cohort Based on ctDNA
Description: pCR and Objective response rate according to RECIST 1.1 per investigator assessment after 24 weeks of treatment
Time Frame: After 24 weeks of treatment
Population: The Full Analysis Set (FAS) comprised all randomized participants in the study. This analysis was to be done in PIK3CA wild-type patients based on Circulating tumor DNA (ctDNA). Data could not be reported in this table as the ctDNA analysis was not done after the primary endpoint was negative.
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Rate of Breast Conserving Surgery for Alpelisib vs. Placebo - PIK3CA Mutant Cohort
Description: Breast conserving surgery is defined for participants who underwent surgery and did not have a mastectomy. The row "no surgery" provides the number of patients who did not undergo surgery at all for various reasons.
Time Frame: After 24 weeks of treatment
Population: The Full Analysis Set (FAS) for the PIK3CA mutant cohort comprised all randomized participants who were assigned to the PIK3CA mutant cohort based on tumor tissue for the randomization. PIK3CA mutation is based on tumor tissue.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 60 | 67
Percentage of participants
  Breast conserving surgery | 56.7 [47.6 to 65.4] | 50.7 [42.2 to 59.2]
  No Surgery | 15.0 [9.3 to 22.6] | 9.0 [4.8 to 15.2]

8. Secondary Outcome: Rate of Breast Conserving Surgery for Alpelisib vs. Placebo - PIK3CA Wild-type Cohort
Description: Breast conserving surgery is defined as the percentage of participants with no mastectomy following completion of 24 weeks of treatment. Breast conserving surgery is defined for participants who underwent surgery and did not have a mastectomy. The row "no surgery" provides the number of patients who did not undergo surgery at all for various reasons.
Time Frame: After 24 weeks of treatment
Population: The Full Analysis Set (FAS) for the PIK3CA wild-type cohort comprised all randomized participants who were assigned to the PIK3CA wild-type cohort based on tumor tissue for the randomization. PIK3CA mutation is based on tumor tissue.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 71 | 59
Percentage of participants
  Breast conserving surgery | 50.7 [42.5 to 58.9] | 62.7 [53.6 to 71.2]
  No Surgery | 18.3 [12.5 to 25.6] | 8.5 [4.5 to 15.2]

9. Secondary Outcome: Association Between pCR and Changes in Ki67 From Baseline for Alpelisib vs. Placebo - PIK3CA Mutant Cohort: Responders as Per pCR
Description: Association Between pCR and Changes in Ki67 From Baseline for Alpelisib vs. Placebo - PIK3CA Mutant Cohort: Responders as Per pCR
Time Frame: Baseline, Cycle 1 Day 15 (each cycle is 28 days) and surgery (End of Treatment (EOT) expected after 24 weeks of treatment)
Population: The FAS for the PIK3CA mutant cohort comprised all randomized participants who were assigned to the PIK3CA mutant cohort based on tumor tissue for the randomization. Only responders as per pCR were considered for this analysis. No patient had data reported at end of trial (EOT), hence the percent change from baseline at EOT could not be reported.
Measure: Median (Full Range); unit: Percentage of positive cells
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 1 | 2
Percentage of positive cells
  Baseline | 5.0 [5 to 5] | 11.0 [5 to 17]
  C1D15: % change from Baseline: number analyzed (Participants) | 1 | 1
  C1D15: % change from Baseline | -80.0 [-80 to -80] | 80.0 [80 to 80]
  EOT % change from Baseline: number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Association Between pCR and Changes in Ki67 From Baseline for Alpelisib vs. Placebo - PIK3CA Mutant Cohort: Non-responders as Per pCR
Description: Association Between pCR and Changes in Ki67 From Baseline for Alpelisib vs. Placebo - PIK3CA Mutant Cohort: Non-responders as Per pCR.
Time Frame: Baseline, Cycle 1 Day 15 (each cycle is 28 days ) and surgery (End of Treatment (EOT) expected after 24 weeks of treatment)
Population: The Full Analysis Set (FAS) for the PIK3CA mutant cohort comprised all randomized participants who were assigned to the PIK3CA mutant cohort based on tumor tissue for the randomization. Only non-responders as per pCR are considered for this analysis.
Measure: Median (Full Range); unit: Percentage of positive cells
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 59 | 65
Percentage of positive cells
  Baseline | 14.0 [0 to 82] | 13.0 [3 to 89]
  C1D15 % change from Baseline: number analyzed (Participants) | 45 | 52
  C1D15 % change from Baseline | -62.5 [-97 to 467] | -60.0 [-96 to 733]
  EOT % change from Baseline: number analyzed (Participants) | 34 | 49
  EOT % change from Baseline | -51.2 [-94 to 400] | -60.0 [-97 to 223]

11. Secondary Outcome: Association Between pCR and Changes in Ki67 From Baseline for Alpelisib vs. Placebo - PIK3CA Wild-type Cohort: Responders as Per pCR
Description: Association between pCR and changes in Ki67 from baseline for alpelisib vs. placebo - PIK3CA wild-type cohort: responders as per pCR
Time Frame: as for outcome 9
Population: FAS for PIK3CA wild-type cohort comprised all rand. Parts. assigned to PIK3CA wild-type cohort based on tumor tissue for rand. Only responders as per pCR were considered for this analysis. No patient had data reported at C1D15 & EOT for Placebo, hence percent change from baseline could not be reported.
Measure: Median (Full Range); unit: Percentage of positive cells
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 2 | 1
Percentage of positive cells
  Baseline | 16.5 [3 to 30] | 20.0 [20 to 20]
  C1D15: % change from Baseline: number analyzed (Participants) | 1 | 0
  C1D15: % change from Baseline | -80.0 [-80 to -80] |
  EOT % change from Baseline: number analyzed (Participants) | 2 | 0
  EOT % change from Baseline | -45.0 [-90 to 0] |

12. Secondary Outcome: Association Between pCR and Changes in Ki67 From Baseline for Alpelisib vs. Placebo - PIK3CA Wild-type Cohort: Non-responders as Per pCR
Description: Association between pCR and changes in Ki67 from baseline for alpelisib vs. placebo - PIK3CA wild-type cohort: non-responders as per pCR
Time Frame: as for outcome 9
Population: The Full Analysis Set (FAS) for the PIK3CA wild-type cohort comprised all randomized participants who were assigned to the PIK3CA wild-type cohort based on tumor tissue for the randomization. Only non-responders as per pCR are considered for this analysis.
Measure: Median (Full Range); unit: Percentage of positive cells
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 69 | 58
Percentage of positive cells
  Baseline | 16.0 [3 to 60] | 18.0 [4 to 85]
  C1D15 % change from Baseline: number analyzed (Participants) | 51 | 47
  C1D15 % change from Baseline | -60.0 [-97 to 220] | -52.0 [-93 to 50]
  EOT % change from Baseline: number analyzed (Participants) | 37 | 41
  EOT % change from Baseline | -60.0 [-90 to 190] | -71.1 [-100 to 250]

13. Secondary Outcome: Preoperative Endocrine Prognostic Index (PEPI) Response as Per Central Assessment for Alpelisib vs. Placebo - PIK3CA Mutant Cohort
Description: Preoperative endocrine prognostic index (PEPI) response as per central assessment for alpelisib vs. placebo - PIK3CA mutant cohort. The total PEPI score assigned to each patient is the sum of the risk points derived from the pT stage, pN stage, Ki67 level, and ER status of the surgical specimen (Ellis et al, Contemp Clin Trials 2008). The PEPI score ranges from 0 to to 12, and a higher score means a worse outcome. PEPI response is defined as a PEPI score of 0.
Time Frame: At the time of surgery (expected after 24 weeks of treatment)
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 60 | 67
Number of participants | 1 | 0

14. Secondary Outcome: Preoperative Endocrine Prognostic Index (PEPI) Response as Per Central Assessment for Alpelisib vs. Placebo - PIK3CA Wild-type Cohort
Description: Preoperative endocrine prognostic index (PEPI) response as per central assessment for alpelisib vs. placebo - PIK3CA wild-type cohort. The total PEPI score assigned to each patient is the sum of the risk points derived from the pT stage, pN stage, Ki67 level, and ER status of the surgical specimen (Ellis et al, Contemp Clin Trials 2008). The PEPI score ranges from 0 to to 12, and a higher score means a worse outcome. PEPI response is defined as a PEPI score of 0.
Time Frame: At the time of surgery (expected after 24 weeks of treatment)
Population: as for outcome 2
Measure: Number; unit: Number of participants
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 71 | 59
Number of participants | 1 | 1

15. Secondary Outcome: Alpelisib PK Parameters: AUC0-24, AUClast at Cycle 1 Day 1
Description: Summary of primary PK parameters for alpelisib plasma concentration
Time Frame: 0, 0.5, 1, 3, 6, 9 and 24 hours post-dose at Cycle 1 Day 1 (each cycle is 28 days)
Population: The BYL FPAS included participants who received at least 1 dose of alpelisib, had at least 1 evaluable post-treatment alpelisib concentration, received adequate doses of alpelisib and letrozole prior to full PK assessment, did not vomit within 4 hours of alpelisib or letrozole dosing on the day of full PK and had an evaluable full PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Alpelisib + Letrozole
Number analyzed (Participants) | 5
ng*hr/mL
  AUC0-24: number analyzed (Participants) | 3
  AUC0-24 | 30800 (20.6)
  AUClast | 27300 (68.6)

16. Secondary Outcome: Alpelisib PK Parameter: Cmax at Cycle 1 Day 1
Description: Summary of primary PK parameters for alpelisib plasma concentration
Time Frame: Cycle 1 Day 1 (each cycle is 28 days)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alpelisib + Letrozole
Number analyzed (Participants) | 5
ng/mL | 3160 (25.3)

17. Secondary Outcome: Alpelisib and PK Parameter: Tmax at Cycle 1 Day 1
Description: Summary of primary PK parameters for alpelisib plasma concentration
Time Frame: Cycle 1 Day 1 (each cycle is 28 days)
Population: Alpelisib Pharmacokinetic Analysis Set (BYL PAS): The BYL PAS included all participants who received at least one dose of alpelisib and had at least one evaluable post-treatment alpelisib concentration measurement.
Measure: Median (Full Range); unit: HR
Arm/Group | Alpelisib + Letrozole
Number analyzed (Participants) | 5
HR | 2.93 [1 to 6]

18. Secondary Outcome: Alpelisib PK Parameters: AUC0-24, AUClast at Cycle 4 Day 1
Description: Summary of primary PK parameters for alpelisib plasma concentration
Time Frame: 0, 0.5, 1, 3, 6, 9 and 24 hours post-dose at Cycle 4 Day 1 (each cycle is 28 days)
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Alpelisib + Letrozole
Number analyzed (Participants) | 5
ng*hr/mL
  AUC0-24: number analyzed (Participants) | 2
  AUC0-24 | 38000 (13.2)
  AUClast: number analyzed (Participants) | 2
  AUClast | 38000 (13.1)

19. Secondary Outcome: Alpelisib PK Parameter: Cmax at Cycle 4 Day 1
Description: Summary of primary PK parameters for alpelisib plasma concentration
Time Frame: Cycle 4 Day 1 (each cycle is 28 days)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alpelisib + Letrozole
Number analyzed (Participants) | 5
ng/mL | 3260 (26.7)

20. Secondary Outcome: Alpelisib PK Parameter: Tmax at Cycle 4 Day 1
Description: Summary of primary PK parameters for alpelisib plasma concentration
Time Frame: Cycle 4 Day 1 (each cycle is 28 days)
Population: as for outcome 17
Measure: Median (Full Range); unit: hr
Arm/Group | Alpelisib + Letrozole
Number analyzed (Participants) | 5
hr | 2.99 [2.98 to 3]

21. Secondary Outcome: Letrozole and PK Parameters: AUC0-24, AUClast at Cycle 1 Day 1
Description: Summary of primary PK parameters for Letrozole plasma concentration
Time Frame: 0, 0.5, 1, 3, 6, 9 and 24 hours post-dose at Cycle 1 Day 1 (each cycle is 28 days)
Population: The LZ FPAS included participants who received at least 1 dose of letrozole, had at least 1 evaluable post-treatment letrozole concentration, received adequate doses of letrozole prior to full PK assessment, did not vomit within 4 hours of letrozole dosing on the day of full PK and had an evaluable full PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 5 | 15
ng*hr/mL
  AUC0-24: number analyzed (Participants) | 3 | 10
  AUC0-24 | 433 (36.3) | 427 (28.8)
  AUClast: number analyzed (Participants) | 5 | 14
  AUClast | 314 (96.9) | 347 (49.6)

22. Secondary Outcome: Letrozole PK Parameter: Cmax at Cycle 1 Day 1
Description: Summary of primary PK parameters for letrozole plasma concentration
Time Frame: Cycle 1 Day 1 (each cycle is 28 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 5 | 15
ng/mL | 30.2 (33.2) | 28 (42.3)

23. Secondary Outcome: Letrozole PK Parameter: Tmax at Cycle 1 Day 1
Description: Summary of primary PK parameters for letrozole plasma concentration
Time Frame: Cycle 1 Day 1 (each cycle is 28 days)
Population: as for outcome 21
Measure: Median (Full Range); unit: hr
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 5 | 15
hr | 1.03 [1 to 3] | 2.25 [1 to 24.5]

24. Secondary Outcome: Letrozole PK Parameters: AUC0-24, AUClast at Cycle 4 Day 1
Description: Summary of primary PK parameters for Letrozole plasma concentration
Time Frame: 0, 0.5, 1, 3, 6, 9 and 24 hours post-dose at Cycle 4 Day 1 (each cycle is 28 days)
Population: Letrozole Pharmacokinetic Analysis Set (LZ PAS): The LZ PAS included all participants who received at least one dose of letrozole and had at least one evaluable post-treatment letrozole concentration measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 5 | 15
ng*hr/mL
  AUC0-24: number analyzed (Participants) | 2 | 8
  AUC0-24 | 1280 (18) | 1810 (33.1)
  AUClast: number analyzed (Participants) | 2 | 13
  AUClast | 1280 (17.9) | 1440 (66.7)

25. Secondary Outcome: Letrozole PK Parameter: Cmax at Cycle 4 Day 1
Description: Summary of primary PK parameters for letrozole plasma concentration
Time Frame: Cycle 4 Day 1 (each cycle is 28 days)
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 5 | 15
ng/mL | 75.6 (6.84) | 103 (30)

26. Secondary Outcome: Letrozole PK Parameter: Tmax at Cycle 4 Day 1
Description: Summary of primary PK parameters for letrozole plasma concentration
Time Frame: Cycle 4 Day 1 (each cycle is 28 days)
Population: as for outcome 21
Measure: Median (Full Range); unit: hr
Arm/Group | Alpelisib + Letrozole | Placebo + Letrozole
Number analyzed (Participants) | 5 | 15
hr | 2 [1 to 3] | 1.17 [1 to 6]

27. Secondary Outcome: Buparlisib PK Parameters: AUC0-24, AUClast at Cycle 1 Day 1
Description: Summary of primary PK parameters for Buparlisib plasma concentration
Time Frame: 0, 0.5, 1, 3, 6, 9 and 24 hours post-dose at Cycle 1 Day 1 (each cycle is 28 days)
Population: The BKM FPAS included participants who received at least 1 dose of buparlisib, had at least 1 evaluable post-treatment concentration, received adequate doses of buparlisib and letrozole prior to full PK assessment, did not vomit within 4 hours of buparlisib or letrozole dosing on the day of full PK and had an evaluable full PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Buparlisib + Letrozole
Number analyzed (Participants) | 10
ng*hr/mL
  AUC0-24: number analyzed (Participants) | 8
  AUC0-24 | 6420 (60)
  AUClast: number analyzed (Participants) | 9
  AUClast | 4820 (123)

28. Secondary Outcome: Buparlisib PK Parameter: Cmax at Cycle 1 Day 1
Description: Summary of primary PK parameters for buparlisib plasma concentration
Time Frame: Cycle 1 Day 1 (each cycle is 28 days)
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Buparlisib + Letrozole
Number analyzed (Participants) | 10
ng/mL | 760 (86.7)

29. Secondary Outcome: Buparlisib PK Parameter: Tmax at Cycle 1 Day 1
Description: Summary of primary PK parameters for buparlisib plasma concentration
Time Frame: Cycle 1 Day 1 (each cycle is 28 days)
Population: Buparlisib Pharmacokinetic Analysis Set (BKM PAS): The BKM PAS included all participants who received at least one dose of buparlisib and had at least one evaluable post-treatment buparlisib concentration measurement.
Measure: Median (Full Range); unit: hr
Arm/Group | Buparlisib + Letrozole
Number analyzed (Participants) | 10
hr | 1.03 [0.5 to 3.5]

30. Secondary Outcome: Buparlisib PK Parameter: AUClast at Cycle 4 Day 1
Description: Summary of primary PK parameters for Buparlisib plasma concentration
Time Frame: 0, 0.5, 1, 3, 6, 9 and 24 hours post-dose at Cycle 4 Day 1 (each cycle is 28 days)
Population: BKM FPAS: The BKM FPAS included participants who received at least 1 dose of buparlisib, had at least 1 evaluable post-treatment concentration, received adequate doses of buparlisib and letrozole prior to full PK assessment, did not vomit within 4 hours of buparlisib or letrozole dosing on the day of full PK and had an evaluable full PK profile.
Measure: Median (Full Range); unit: ng*hr/mL
Arm/Group | Buparlisib + Letrozole
Number analyzed (Participants) | 10
ng*hr/mL | 10400 [10400 to 10400]

31. Secondary Outcome: Buparlisb PK Parameter: Cmax at Cycle 4 Day 1
Description: Summary of primary PK parameters for buparlisib plasma concentration
Time Frame: Cycle 4 Day 1 (each cycle is 28 days)
Population: as for outcome 29
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Buparlisib + Letrozole
Number analyzed (Participants) | 10
ng/mL | 610 [610 to 610]

32. Secondary Outcome: Buparlisib PK Parameter: Tmax at Cycle 4 Day 1
Description: Summary of primary PK parameters for buparlisib plasma concentration
Time Frame: Cycle 4 Day 1 (each cycle is 28 days)
Population: as for outcome 29
Measure: Median (Full Range); unit: hr
Arm/Group | Buparlisib + Letrozole
Number analyzed (Participants) | 10
hr | 3 [3 to 3]

ADVERSE EVENTS:
Time Frame: All Adverse Events reported in this record are on-treatment events (from first dose of study treatment to last dose of study treatment + 30 days, duration expected to be a total of approximately 25 weeks).
Description: Adverse Events, Serious Adverse Events based on Safety Set population defined as all patients who received at least one dose of study treatment
Arm/Group | Alpelisib + Letrozole | Buparlisib + Letrozole | Placebo + Letrozole
All-Cause Mortality (participants affected / at risk) | 1/130 | 0/81 | 1/125
Serious Adverse Events (participants affected / at risk) | 21/130 | 22/81 | 6/125
Other Adverse Events (participants affected / at risk) | 126/130 | 80/81 | 106/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpelisib + Letrozole (N=130) | Buparlisib + Letrozole (N=81) | Placebo + Letrozole (N=125)
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Iritis (Eye disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 2 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 3 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 7 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 6 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alpelisib + Letrozole (N=130) | Buparlisib + Letrozole (N=81) | Placebo + Letrozole (N=125)
Tachycardia (Cardiac disorders) | 3 | 5 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 5 | 6
Vision blurred (Eye disorders) | 9 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 6 | 4
Abdominal pain (Gastrointestinal disorders) | 7 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7 | 4
Constipation (Gastrointestinal disorders) | 5 | 7 | 13
Diarrhoea (Gastrointestinal disorders) | 66 | 29 | 19
Dry mouth (Gastrointestinal disorders) | 14 | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 11 | 11 | 6
Nausea (Gastrointestinal disorders) | 57 | 37 | 23
Stomatitis (Gastrointestinal disorders) | 42 | 18 | 5
Vomiting (Gastrointestinal disorders) | 23 | 6 | 6
Asthenia (General disorders) | 21 | 16 | 17
Chills (General disorders) | 7 | 8 | 5
Fatigue (General disorders) | 53 | 30 | 42
Mucosal dryness (General disorders) | 7 | 2 | 0
Oedema peripheral (General disorders) | 9 | 4 | 4
Pyrexia (General disorders) | 12 | 1 | 3
Urinary tract infection (Infections and infestations) | 15 | 7 | 7
Viral upper respiratory tract infection (Infections and infestations) | 5 | 5 | 13
Procedural pain (Injury, poisoning and procedural complications) | 2 | 5 | 9
Alanine aminotransferase increased (Investigations) | 14 | 49 | 3
Aspartate aminotransferase increased (Investigations) | 11 | 44 | 2
Blood bilirubin increased (Investigations) | 2 | 6 | 1
Blood creatinine increased (Investigations) | 12 | 1 | 4
Blood glucose increased (Investigations) | 12 | 3 | 2
Gamma-glutamyltransferase increased (Investigations) | 5 | 6 | 1
Weight decreased (Investigations) | 16 | 10 | 3
Decreased appetite (Metabolism and nutrition disorders) | 40 | 25 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 69 | 38 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 13 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 5 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 13
Dizziness (Nervous system disorders) | 7 | 22 | 19
Dysgeusia (Nervous system disorders) | 24 | 11 | 7
Headache (Nervous system disorders) | 26 | 10 | 16
Memory impairment (Nervous system disorders) | 2 | 5 | 2
Paraesthesia (Nervous system disorders) | 8 | 2 | 4
Tremor (Nervous system disorders) | 0 | 8 | 1
Anxiety (Psychiatric disorders) | 10 | 16 | 10
Depression (Psychiatric disorders) | 5 | 12 | 3
Insomnia (Psychiatric disorders) | 15 | 8 | 17
Breast pain (Reproductive system and breast disorders) | 4 | 8 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 3 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 19 | 14 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 18 | 9
Rash (Skin and subcutaneous tissue disorders) | 58 | 31 | 10
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22 | 9 | 3
Hot flush (Vascular disorders) | 8 | 12 | 31
Hypertension (Vascular disorders) | 16 | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT01923168/SAP_000.pdf
  • Study Protocol (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT01923168/Prot_001.pdf